CLINICAL TRIAL: NCT00682877
Title: A Comparison Trial of SmartPill Corporation GI Monitoring System With Scintigraphic Gastric Emptying Procedure for Determining Gastric Residence Time - In Subjects Over 65 Years of Age
Brief Title: A Comparison of SmartPill Capsule With Scintigraphy for Determining Gastric Residence Time - Over 65 Years Old
Acronym: GETOver65
Status: Completed | Type: Observational
Sponsor: The SmartPill Corporation (Industry)
Responsible Party: John R. Semler/Chief Technology Officer, The SmartPill Corporation
Other Study IDs: 102204a
Record Dates: First submitted 2008-05-20; First posted 2008-05-23 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Gastrointestinal Diseases; Stomach Diseases; Gastroparesis
Keywords: gastroparesis; Digestive; Gastrointestinal; Stomach; Motility; Non-Invasive; Capsule; GI; Device; Digestive System Diseases
MeSH Terms: conditions — Gastrointestinal Diseases; Stomach Diseases; Gastroparesis; Digestive System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: healthy adult subjects with no history or current gastrointestinal disorders or conditions
- Gastroparesis: Subjects with documented gastroparesis

SUMMARY:
The purpose of this study is to determine the correlation between gastric residence time of the SmartPill Capsule and the time required for partial emptying of a standard radiolabeled meal as measured by gastric emptying scintigraphy for subjects 65 years of age and older.

DETAILED DESCRIPTION:
Gastric emptying scintigraphy is considered the gold standard for evaluating gastric emptying and is widely available. Accurate characterization of gastric emptying may guide medical and surgical treatment choices. In addition, these techniques may allow for monitoring of therapeutic results for follow-up patient management.

The SmartPill GI Monitoring System offers an alternative non-invasive method for characterizing disorders of the stomach. The system consists of an ingestible capsule that houses sensors for pH, temperature, and pressure, a receiver for receiving and storing signals from the capsule, and software for displaying data on a personal computer. The capsule samples at regular intervals and transmits the sensed pH, pressure, and temperature data to a portable receiver worn by the subject. After test completion, the recorded data is downloaded to a personal computer for subsequent evaluation. This trial is for subjects 65 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria For Healthy Subjects:

  * Healthy males and females between ages 65-80 years of age with no gastrointestinal disease as screened by the GI Disease Screening Questionnaire
  * Average bowel movement frequency of at least one bowel movement within 48 hours
  * Subjects with high probability for compliance and completion of the study
* Inclusion Criteria For Subjects with Gastroparesis:

  * Abnormal gastric emptying as defined by local standards and documented by nuclear medicine scintigraphy performed within the last two years.
  * Males and females between ages 18-65 years of age.
  * Average bowel movement frequency of at least one bowel movement within 72 hours
  * Subjects with high probability for compliance and completion of the study
  * Upper endoscopy or upper GI within last 3 years showing no evidence of gastric bezoar, stricture, or peptic ulcer.

Exclusion Criteria:

* Exclusion Criteria For Healthy Subjects:

  * Prior GI surgery
  * Surgery within the past 3 months
  * Diverticulitis
  * Tobacco use within eight hours prior to capsule ingestion and during the 8 hour monitoring time.
  * Alcohol use within 24 hours prior to capsule ingestion and throughout the entire monitoring period (up to 72 hours).
  * Body mass index (BMI) > 35
  * Allergies to components of the test meal including eggs, bread, and jam.
  * Female of childbearing age who is not practicing birth control and/or is pregnant or lactating. (Confirm with urine pregnancy test)
  * Cardiovascular, endocrine, renal, or other chronic disease likely to affect motility.
* Exclusion Criteria For Subjects with Gastroparesis:

  * History of gastric bezoar
  * Severe dysphagia to solid food and pills
  * Severe vomiting more than 1 time per day
  * Diverticulitis
  * Severe daily abdominal pain requiring medications for relief
  * Severe weight loss, greater than 10 lbs over the preceding 2 months.
  * Uncontrolled diabetes with a hemoglobin A1C greater than 10.
  * Excessively delayed gastric emptying time: more than 90% of a standard egg meal retained after 2 hours.
  * Previous gastro-esophageal surgery including vagotomy, fundoplication, gastric bypass, ulcer surgery.
  * Prior GI surgery except for uncomplicated appendectomy and laparoscopic cholecystectomy
  * Surgery within the past 3 months
  * Tobacco use within eight hours prior to capsule ingestion and during the 8 hour monitoring time.
  * Alcohol use within 24 hours prior to capsule ingestion and throughout the entire monitoring period (up to 72 hours).
  * BMI > 35
  * Allergies to components of the test meal including eggs, bread, and jam
  * Female of childbearing age who is not practicing birth control and/or is pregnant or lactating. (Confirm with urine pregnancy test)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: patients with gastroparesis referred to a tertiary motility center - 65 years of age and older.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-07; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To demonstrate the correlation between the gastric residence time as determined by SmartPill GI Monitoring System and the gastric emptying time of a radiolabeled meal in both healthy subjects and patients with documented gastroparesis. | 30 minute intervals up to 6 hours

SECONDARY OUTCOMES:
To demonstrate that the gastric residence time as determined by SmartPill GI Monitoring System can discriminate between healthy human subjects and patients with gastroparesis | Continuous time measure until capsule elimination
To characterize pressure patterns within the antrum and duodenum in healthy subjects and patients with documented gastroparesis | Continuous time measure until capsule elimination
To characterize total GI transit time in healthy subjects | Continuous time measure until capsule elimination

CONTACTS AND LOCATIONS:
Overall Officials: Braden Kuo, MD, Principal Investigator — Massachusetts General Hospital; John R Semler, PhD, Study Director — SmartPill Corporation
Locations (2):
- United States (2):
  - Division of Gastroenterology and Hepatology at KUMC, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts